CLINICAL TRIAL: NCT00320541
Title: A Randomized Phase II Trial of Paclitaxel and Bevacizumab Versus Gemcitabine, Paclitaxel, and Bevacizumab as First Line Treatment for Locally Advanced or Metastatic Breast Cancer
Brief Title: A Trial of Paclitaxel and Bevacizumab vs. Gemcitabine, Paclitaxel, and Bevacizumab in Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10663; B9E-US-S377 (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Results first posted 2010-07-27 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Cancer of Breast; Cancer of the breast; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- paclitaxel plus bevacizumab (PB) (Active Comparator): paclitaxel 90 milligrams per meter squared (mg/m2) administered intravenously (IV) on days 1, 8, 15 every 28 days followed by bevacizumab 10 milligrams per kilogram (mg/kg) administered IV on days 1 and 15 every 28 days
  Interventions: Drug: paclitaxel; Drug: bevacizumab
- paclitaxel plus bevacizumab plus gemcitabine (PB+G) (Experimental): paclitaxel 90 milligrams per meter squared (mg/m2) administered intravenously (IV) on days 1, 8, 15 every 28 days followed by gemcitabine 1500 mg/m2 IV on days 1 and 15 every 28 days followed by bevacizumab 10 milligrams per kilogram (mg/kg) administered IV on days 1 and 15 every 28 days
  Interventions: Drug: gemcitabine; Drug: paclitaxel; Drug: bevacizumab

INTERVENTIONS:
Drug: gemcitabine — 1500 mg/m2, IV day 1 and day 15 every 28 days until complete response, disease progression or unacceptable toxicity
  Other Names: LY188011; Gemzar
  Arms: paclitaxel plus bevacizumab plus gemcitabine (PB+G)
Drug: paclitaxel — 90 mg/m2, IV, day 1, day 8 and day 15 every 28 days until complete response, disease progression or unacceptable toxicity
  Other Names: Taxol
Drug: bevacizumab — 10 mg/kg, IV, day 1 and day 15 every 28 days until complete response, disease progression or unacceptable toxicity
  Other Names: Avastin

SUMMARY:
This study will compare the cancer response to both treatments for locally advanced or metastatic breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Females diagnosed with breast cancer and the cancer has spread to distant areas of the breast or organs.
* Must be able to measure the disease by specific medical parameters
* May have received breast cancer treatment in the early stage of the disease
* May be restricted in physically strenuous activity but able to carry out light work.
* Must have adequate organ function as seen in blood test results.

Exclusion

Criteria:

* Cancer that has spread to the brain.
* Unstable heart problems
* Unstable high blood pressure.
* Breast cancer treatment after the disease has considered to spread to other areas or organs.
* Unable to agree with the requirements of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2006-05; Primary Completion 2009-04 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (32):
- United States (30):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fayetteville, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Jolla, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mission Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Rosa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Muncie, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Southfield, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chesterfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Missoula, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Akron, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dayton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dunmore, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lubbock, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Everett, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milwaukee, Wisconsin
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 219 patients were screened; 28 patients were screen failures and were not assigned treatment.
Period: Overall Study
Arm/Group | Paclitaxel Plus Bevacizumab (PB) | Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G)
Started | 94 | 93
Completed | 44 | 36
Not Completed | 50 | 57
Not completed — Adverse Event | 21 | 19
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 12 | 16
Not completed — Physician Decision | 9 | 13
Not completed — Other | 3 | 4
Not completed — Sponsor Decision | 2 | 1
Not completed — Death due to Study Disease | 1 | 3
Not completed — Death due to Adverse Event(s) | 1 | 0
Not completed — Protocol Entry Criterion Not Met | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel Plus Bevacizumab (PB) | Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G) | Total
Number analyzed (Participants) | 94 | 93 | 187
Age Continuous [Mean (Standard Deviation); unit: years] | 57.5 (10.68) | 56.8 (9.56) | 57.2 (10.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 93 | 187
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 80 | 77 | 157
  African | 5 | 11 | 16
  Hispanic | 7 | 4 | 11
  East Asian | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 94 | 93 | 187
Basis for Pathological Diagnosis [Number; unit: participants] — Methodology used for obtaining pathological diagnosis
  participants
    Histopathological | 84 | 84 | 168
    Cytological | 10 | 8 | 18
    Missing | 0 | 1 | 1
Breakdown According to Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG Performance Status classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death). In this study, ECOG performance status was assessed within 14 days of Visit 1. Patients were required to have a baseline ECOG Performance Status of 0 or 1 for study participation.
  participants
    Fully Active- 0 | 57 | 60 | 117
    Ambulatory, Restricted Strenuous Activity- 1 | 37 | 31 | 68
    Missing | 0 | 2 | 2
Breakdown by Estrogen Receptor (ER) Status [Number; unit: participants] — Breakdown of participants by ER status
  participants
    Positive | 60 | 67 | 127
    Negative | 33 | 25 | 58
    Unknown | 1 | 1 | 2
Breakdown by Human Epidermal Growth Factor (HER-2 NEU) Status [Number; unit: participants] — Breakdown of participants by HER-2 NEU status
  participants
    Not done | 3 | 4 | 7
    Positive | 4 | 2 | 6
    Negative | 87 | 86 | 173
    Missing | 0 | 1 | 1
Breakdown by Progesterone Receptor (PR) Status [Number; unit: participants] — Breakdown of participants by PR status
  participants
    Not done | 1 | 0 | 1
    Positive | 42 | 57 | 99
    Negative | 50 | 35 | 85
    Unknown | 1 | 1 | 2
Breakdown of Disease-free Interval [Number; unit: participants] — Breakdown by treatment arm of disease-free interval which was defined as the duration between prior adjuvant chemotherapy stop date and disease recurrence date for applicable participants who received adjuvant chemotherapy.
  participants
    Less than or equal to 24 months | 5 | 10 | 15
    Greater than 24 months | 6 | 2 | 8
    Not applicable | 83 | 81 | 164
Diagnosis by pathology [Number; unit: participants] — Pathology of breast cancer diagnosis
  participants
    Ductal breast carcinoma | 76 | 79 | 155
    Lobal breast carcinoma | 9 | 6 | 15
    Tubal breast carcinoma | 0 | 0 | 0
    Medullary breast carcinoma | 0 | 0 | 0
    Adenocystic breast carcinoma | 0 | 0 | 0
    Papillar breast carcinoma | 0 | 0 | 0
    Breast carcinoma | 6 | 3 | 9
    Other | 3 | 5 | 8
Menopausal Status [Number; unit: participants] — Breakdown of menopausal status
  participants
    Not done | 1 | 1 | 2
    Pre-menopausal | 18 | 18 | 36
    Peri-menopausal | 2 | 3 | 5
    Post-menopausal | 73 | 70 | 143
    Unknown | 0 | 1 | 1
Presence of Visceral Metastases [Number; unit: participants] — Presence of visceral metastases at baseline visit
  participants
    Yes | 68 | 66 | 134
    No | 25 | 24 | 49
    Missing | 1 | 3 | 4
Prior Biological Treatment for This Cancer [Number; unit: participants] — Number of participants, by treatment arm, who had received prior biological treatment for this cancer. NOTE: The total number of participants who received prior biological treatment does not equal the total number of participants in the trial because not all participants received prior biological treatment.
  participants | 0 | 2 | 2
Prior Cancer Surgery [Number; unit: participants] — Number of participants, by treatment arm, who underwent prior surgery. NOTE: The total number of participants who underwent prior surgery does not equal the total number of participants in the trial because not all participants underwent prior surgery.
  participants | 79 | 82 | 161
Prior Chemotherapy for This Cancer [Number; unit: participants] — Number of participants, by treatment arm, who received prior chemotherapy for this cancer. NOTE: The total number of participants who received prior chemotherapy does not equal the total number of participants in the trial because not all participants received prior chemotherapy.
  participants | 55 | 57 | 112
Prior Exposure to Taxanes [Number; unit: participants] — Number of participants previously treated with taxane chemotherapy including: Taxol (paclitaxel), Topotecan (docetaxel), or Abraxane (albumin-bound paclitaxel).
  participants
    Yes | 33 | 32 | 65
    No | 61 | 61 | 122
Prior Hormonal Treatment for This Cancer [Number; unit: participants] — Number of participants, by treatment arm, who received prior hormonal treatment for this cancer. NOTE: The total number of participants who received prior hormonal treatment does not equal the total number of participants in the trial because not all participants received prior hormonal treatment.
  participants | 51 | 53 | 104
Prior Immunological Treatment for This Cancer [Number; unit: participants] — Number of participants, by treatment arm, who received prior immunological treatment for this cancer. NOTE: The total number of participants who received prior immunnological treatment does not equal the total number of participants in the trial because not all participants received prior immunological treatment.
  participants | 2 | 0 | 2
Prior Radiotherapy [Number; unit: participants] — Number of participants, by treatment arm, who received prior radiotherapy. NOTE: The total number of participants who received prior radiotherapy does not equal the total number of participants in the trial because not all participants received prior radiotherapy.
  participants | 50 | 55 | 105
Body Surface Area (BSA) at Day 1 of Visit 1 [Mean (Standard Deviation); unit: square meters (m2)] | 1.8 (0.18) | 1.8 (0.21) | 1.8 (0.20)

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Response defined per Response Evaluation Criteria In Solid Tumors (RECIST) criteria: Complete Response (CR)=disappearance of all target lesions; Partial Response (PR)=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that do not meet above criteria. ORR was defined as the proportion of participants who achieved a best response of either CR or PR. ORR=number of participants with CR or PR/number of participants qualified for tumor response analysis (per-protocol population).
Time Frame: baseline & every 2 cycles (approximately 8 weeks) of treatment to measured progressive disease (PD) & post-therapy until PD or other therapy initiated (up to 35 months)
Population: Per-protocol population included intent-to-treat participants who met the following criteria: histological or cytological breast cancer diagnosis; baseline presence of measurable disease per RECIST; at least 1 dose of study drug; no current systemic anti-tumor therapy except protocol-specified therapy. One PB+G participant did not qualify.
Measure: Mean (95% Confidence Interval); unit: proportion of responders
Arm/Group | Paclitaxel Plus Bevacizumab (PB) | Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G)
Number analyzed (Participants) | 94 | 92
proportion of responders | 0.489 [0.385 to 0.595] | 0.587 [0.479 to 0.689]
Statistical Analysis 1: Comparison: Paclitaxel Plus Bevacizumab (PB) vs Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G); Assuming the response rate for the PB arm is 34% and the addition of gemcitabine will improve it to 54%, then a sample size of 170 evaluable participants (85 per arm) will give an 80% statistical power to detect the difference, using a 1-sided test at the significance level of 0.05. Confidence levels are exact binomial 95% Confidence Intervals; Test type: Superiority or Other; p = 0.117, Fisher Exact — Statistical significance at 0.05 level was required

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was measured from date of randomization to first date of disease progression or death from any cause. For participants not known to have died or had disease progression as of data-inclusion cut-off date, PFS duration was censored at date of last study visit prior to data-inclusion cut-off date.
Time Frame: baseline to measured progressive disease or death up to 35 months (tumor assessments were performed every 2 cycles during study therapy; every 2 months during post-therapy until disease progression or new anticancer treatment initiated)
Population: ITT population=all randomized participants, eligible & ineligible. Participants with events: PB=74; PB+G=72. Censored participants: PB=20 PB+G=21.
Measure: Median (Full Range); unit: months
Arm/Group | Paclitaxel Plus Bevacizumab (PB) | Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G)
Number analyzed (Participants) | 94 | 93
months | 8.8 [0.1 to 27.3] | 11.3 [1.5 to 33.8]
Statistical Analysis 1: Comparison: Paclitaxel Plus Bevacizumab (PB) vs Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G); Test type: Superiority or Other; p = 0.247, Log Rank

3. Secondary Outcome: Overall Survival
Description: Overall survival was measured from date of randomization to date of death from any cause. For participants not known to have died as of data-inclusion cut-off date, overall survival duration was censored at date of last study visit prior to the data cut-off date.
Time Frame: baseline to death from any cause (up to 35 months)
Population: Intent-To-Treat (ITT) population=all randomized participants, eligible & ineligible. Number of participants with events: PB=35; PB+G=34. Censored participants: PB=59;PB+G=59.
Measure: Median (Full Range); unit: months
Arm/Group | Paclitaxel Plus Bevacizumab (PB) | Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G)
Number analyzed (Participants) | 94 | 93
months | 25.0 [0.1 to 34.6] | 24.3 [1.5 to 33.8]
Statistical Analysis 1: Comparison: Paclitaxel Plus Bevacizumab (PB) vs Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G); Test type: Superiority or Other; p = 0.475, Log Rank

4. Secondary Outcome: Total Functional Assessment of Cancer Therapy -Breast (FACT-B): Change From Baseline to End of Therapy
Description: FACT-B measures the following domains of health-related quality of life (HR-QL): physical well-being (PWB), social/family well-being (SFWB), emotional well-being (EWB), functional well-being (FWB), & additional concerns of breast cancer (BCS). Total FACT-B scores range from 0-144, with higher scores representing better HR-QOL. Minimally important differences estimates obtained for FACT-B is 7-8 points. FACT-B was assessed at baseline (prior to start of Cycle 1 [Day 1]), prior to start of each subsequent cycle (approximately every 4 weeks) during therapy, through 30-day post therapy follow-up.
Time Frame: Baseline through 30 days post therapy follow-up (up to 35 months)
Population: Last Observation Carried Forward (LOCF) for all ITT patients with valid baseline and at least one valid post-baseline assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paclitaxel Plus Bevacizumab (PB) | Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G)
Number analyzed (Participants) | 60 | 55
units on a scale | -1.0 (15.10) | -10.8 (16.87)
Statistical Analysis 1: Comparison: Paclitaxel Plus Bevacizumab (PB) vs Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G); Test type: Superiority or Other; p = 0.010, ANCOVA; ANCOVA model included treatment arm and baseline assessment

5. Secondary Outcome: Physical Well Being (PWB) Subscale: Change From Baseline to End of Therapy
Description: The PWB subscale of FACT-B measures physical well-being. Total PWB scores range from 0 to 28, with higher scores representing better HR-QOL. FACT-B was assessed at baseline (prior to start of Cycle 1 [Day 1]), then prior to start of each subsequent cycle (approximately every 4 weeks) during therapy, through 30-day post therapy follow-up.
Time Frame: Baseline through 30 days post therapy follow-up (up to 35 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paclitaxel Plus Bevacizumab (PB) | Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G)
Number analyzed (Participants) | 60 | 56
units on a scale | -1.9 (5.90) | -4.0 (6.00)
Statistical Analysis 1: Comparison: Paclitaxel Plus Bevacizumab (PB) vs Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G); Test type: Superiority or Other; p = 0.119, ANCOVA; ANCOVA model included treatment arm and baseline assessment

6. Secondary Outcome: Social/Family Well Being (SFWB) Subscale: Change From Baseline to End of Therapy
Description: The SFWB subscale of FACT-B measures social/family well-being. Total SFWB scores range from 0 to 28, with higher scores representing better HR-QOL. FACT-B was assessed at baseline (prior to start of Cycle 1 [Day 1]), then prior to start of each subsequent cycle (approximately every 4 weeks) during therapy, through 30-day post therapy follow-up.
Time Frame: Baseline through 30 days post therapy follow-up (up to 35 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paclitaxel Plus Bevacizumab (PB) | Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G)
Number analyzed (Participants) | 61 | 56
units on a scale | 0.0 (3.43) | -1.9 (3.61)
Statistical Analysis 1: Comparison: Paclitaxel Plus Bevacizumab (PB) vs Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G); Test type: Superiority or Other; p = 0.023, ANCOVA; ANCOVA model included treatment arm and baseline assessment

7. Secondary Outcome: Emotional Well Being (EWB) Subscale: Change From Baseline to End of Therapy
Description: The EWB subscale of FACT-B measures emotional well-being. Total EWB scores range from 0 to 24, with higher scores representing better HR-QOL. FACT-B was assessed at baseline (prior to start of Cycle 1 [Day 1]), then prior to start of each subsequent cycle (approximately every 4 weeks) during therapy, through 30-day post therapy follow-up.
Time Frame: Baseline through 30 days post therapy follow-up (up to 35 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paclitaxel Plus Bevacizumab (PB) | Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G)
Number analyzed (Participants) | 61 | 56
units on a scale | 1.8 (3.17) | -0.2 (3.88)
Statistical Analysis 1: Comparison: Paclitaxel Plus Bevacizumab (PB) vs Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G); Test type: Superiority or Other; p = 0.002, ANCOVA; ANCOVA model included treatment arm and baseline assessment

8. Secondary Outcome: Functional Well Being (FWB) Subscale: Change From Baseline to End of Therapy
Description: The FWB subscale of FACT-B measures functional well-being. Total FWB scores range from 0 to 28, with higher scores representing better HR-QOL. FACT-B was assessed at baseline (prior to start of Cycle 1 [Day 1]), then prior to start of each subsequent cycle (approximately every 4 weeks) during therapy, through 30-day post therapy follow-up.
Time Frame: Baseline through 30 days post therapy follow-up (up to 35 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paclitaxel Plus Bevacizumab (PB) | Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G)
Number analyzed (Participants) | 61 | 55
units on a scale | -0.3 (5.38) | -3.8 (4.71)
Statistical Analysis 1: Comparison: Paclitaxel Plus Bevacizumab (PB) vs Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G); Test type: Superiority or Other; p = 0.004, ANCOVA; ANCOVA model included treatment arm and baseline assessment

9. Secondary Outcome: Breast Cancer Subscale (BCS): Change From Baseline to End of Therapy
Description: The BCS subscale of FACT-B measures additional concerns of breast cancer . Total BCS scores range from 0 to 36, with higher scores representing better HR-QOL. Minimally important differences estimates obtained for BCS is 2-3 points. FACT-B was assessed at baseline (prior to start of Cycle 1 [Day 1]), then prior to start of each subsequent cycle (approximately every 4 weeks) during therapy, through 30-day post therapy follow-up.
Time Frame: Baseline through 30 days post therapy follow-up (up to 35 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paclitaxel Plus Bevacizumab (PB) | Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G)
Number analyzed (Participants) | 62 | 56
units on a scale | -0.1 (5.02) | -1.9 (4.03)
Statistical Analysis 1: Comparison: Paclitaxel Plus Bevacizumab (PB) vs Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G); Test type: Superiority or Other; p = 0.067, ANCOVA; ANCOVA model included treatment arm and baseline assessment

10. Secondary Outcome: Trial Outcome Index-Breast (TOI-B): Change From Baseline to End of Therapy
Description: The TOI-B represents the total of the subscales PWB,FWB, and BCS. Total TOI-B scores range from 0 to 92, with higher scores representing better HR-QOL. Minimally important differences estimates obtained for TOI is 5-6 points. FACT-B was assessed at baseline (prior to start of Cycle 1 [Day 1]), then prior to start of each subsequent cycle (approximately every 4 weeks) during therapy, through 30-day post therapy follow-up.
Time Frame: Baseline through 30 days post therapy follow-up (up to 35 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paclitaxel Plus Bevacizumab (PB) | Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G)
Number analyzed (Participants) | 60 | 55
units on a scale | -2.5 (12.53) | -9.1 (12.68)
Statistical Analysis 1: Comparison: Paclitaxel Plus Bevacizumab (PB) vs Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G); Test type: Superiority or Other; p = 0.036, ANCOVA; ANCOVA model included treatment arm and baseline assessment

ADVERSE EVENTS:
Description: Adverse events (AEs) provided for all patients who received at least one dose of study drug. AEs are both study-drug related and non-study drug related. AEs represent all grades (1-5). Grade 1: mild adverse event (AE); Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening or disabling AE; Grade 5: death-related to AE.
Arm/Group | Paclitaxel Plus Bevacizumab (PB) | Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G)
Serious Adverse Events (participants affected / at risk) | 27/94 | 36/93
Other Adverse Events (participants affected / at risk) | 93/94 | 93/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel Plus Bevacizumab (PB) (N=94) | Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G) (N=93)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 9 (9)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 3 (3)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 4 (4)
Tenderness (General disorders) | 0 (0) | 1 (1)
Visceral oedema (General disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 5 (7)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (4) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
International normalised ratio (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (6) | 5 (5)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myopathy toxic (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Haemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Central venous catheter removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (2)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Epistaxis (Vascular disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel Plus Bevacizumab (PB) (N=94) | Paclitaxel Plus Bevacizumab Plus Gemcitabine (PB+G) (N=93)
Anaemia (Blood and lymphatic system disorders) | 18 (38) | 35 (76)
Leukopenia (Blood and lymphatic system disorders) | 15 (43) | 23 (82)
Neutropenia (Blood and lymphatic system disorders) | 39 (119) | 65 (169)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (13) | 21 (43)
Tachycardia (Cardiac disorders) | 7 (8) | 6 (6)
Lacrimation increased (Eye disorders) | 6 (6) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 9 (11) | 9 (10)
Constipation (Gastrointestinal disorders) | 29 (38) | 37 (54)
Diarrhoea (Gastrointestinal disorders) | 36 (54) | 47 (58)
Dyspepsia (Gastrointestinal disorders) | 9 (10) | 11 (12)
Haemorrhoids (Gastrointestinal disorders) | 5 (6) | 6 (6)
Nausea (Gastrointestinal disorders) | 40 (59) | 58 (85)
Stomatitis (Gastrointestinal disorders) | 29 (36) | 33 (43)
Vomiting (Gastrointestinal disorders) | 23 (30) | 30 (38)
Asthenia (General disorders) | 12 (13) | 5 (5)
Chills (General disorders) | 5 (5) | 10 (12)
Fatigue (General disorders) | 58 (104) | 74 (129)
Influenza like illness (General disorders) | 2 (2) | 5 (5)
Oedema peripheral (General disorders) | 19 (20) | 24 (32)
Pain (General disorders) | 8 (8) | 12 (13)
Pyrexia (General disorders) | 17 (21) | 25 (33)
Infection (Infections and infestations) | 1 (1) | 5 (6)
Sinusitis (Infections and infestations) | 14 (21) | 13 (13)
Upper respiratory tract infection (Infections and infestations) | 10 (14) | 13 (14)
Urinary tract infection (Infections and infestations) | 18 (25) | 17 (22)
Alanine aminotransferase increased (Investigations) | 2 (2) | 12 (16)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 13 (19)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 5 (7)
Weight decreased (Investigations) | 15 (15) | 16 (22)
Anorexia (Metabolism and nutrition disorders) | 19 (24) | 20 (28)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 8 (14) | 10 (14)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (13) | 7 (12)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (3) | 7 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5) | 6 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 8 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (26) | 20 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (15) | 18 (21)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 14 (18)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 9 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 20 (22) | 15 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (16) | 16 (19)
Dizziness (Nervous system disorders) | 14 (15) | 10 (10)
Dysgeusia (Nervous system disorders) | 9 (10) | 12 (13)
Headache (Nervous system disorders) | 23 (25) | 26 (30)
Neuropathy (Nervous system disorders) | 8 (9) | 10 (13)
Neuropathy peripheral (Nervous system disorders) | 14 (19) | 9 (10)
Paraesthesia (Nervous system disorders) | 5 (6) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 49 (72) | 42 (53)
Anxiety (Psychiatric disorders) | 15 (17) | 9 (11)
Confusional state (Psychiatric disorders) | 0 (0) | 5 (5)
Depression (Psychiatric disorders) | 11 (11) | 8 (8)
Insomnia (Psychiatric disorders) | 13 (16) | 18 (21)
Dysuria (Renal and urinary disorders) | 7 (7) | 5 (5)
Pollakiuria (Renal and urinary disorders) | 5 (5) | 3 (3)
Proteinuria (Renal and urinary disorders) | 3 (11) | 8 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (30) | 25 (36)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 (22) | 25 (29)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 6 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (9)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 10 (11)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 8 (8)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 41 (42) | 44 (49)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 10 (10)
Erythema (Skin and subcutaneous tissue disorders) | 7 (7) | 7 (10)
Nail disorder (Skin and subcutaneous tissue disorders) | 17 (25) | 21 (25)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 18 (23) | 28 (34)
Hot flush (Vascular disorders) | 6 (6) | 7 (9)
Hypertension (Vascular disorders) | 22 (25) | 16 (23)
Epistaxis (Vascular disorders) | 41 (51) | 40 (49)

LIMITATIONS AND CAVEATS:
Of 191 randomized patients, 4 patients were disqualified from inclusion in any efficacy or safety analyses due to significant Good Clinical Practice (GCP) violations; data is reported for the remaining 187 randomized patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days